CLINICAL TRIAL: NCT00987077
Title: Selective Retina Therapy (SRT) in Patients With Idiopathic Central Serous Chorioretinopathy: A Prospective Randomized Controlled Trial
Brief Title: Selective Retina Therapy (SRT) in Patients With Idiopathic Central Serous Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kiel (Other)
Collaborators: Medical Laser Center Lübeck, Lübeck, Germany (Unknown); Institute for Medical Informaties and Statistics Kiel, Germany (Unknown)
Responsible Party: University Eye Clinic Kiel, Germany
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRT_CSC_Kiel
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Central Serous Chorioretinopathy; Selective Retina Therapy
Keywords: CSC; SRT
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Selective Retinatherapy (SRT) (Experimental): Treatment was performed with the SRT-Laser system (Medical Laser Center Lübeck, Germany), which consists of a Q-switched frequency doubled Nd:YLF laser (527nm), operating with a pulse repetition rate of 100 Hz. The pulse duration (full width at half maximum) was 1.7 µs. The laser energy was transmitted via fiber to a Lumenis slitlamp allowing the application of a fixed spot size diameter of 200 µm in air. A Mainster central field contact lens with a magnification of 1.05 was used for all irradiations. Per foot switch, 30 pulses are emitted, the pulse energy was chosen by the physician up to a maximum of 370 µJ. According to the treatment protocol, prior to each treatment 5 test shots with increasing energy were applied adjacent to the vessel arcades, in each patient in order to determine the appropriate pulse energy for treatment by recording the OA-value.
  Interventions: Device: Selective Retina Therapy (SRT)
- control group (No Intervention): Patients randomized to control group achieve no treatment and are followed up for three months.
- crossover (Experimental): After 3 months follow up patients of control group with persistence of disease activity were allocated to crossover group and received either SRT. Crossover group was followed up for further 3 months.
  Interventions: Device: Selective Retina Therapy (SRT)

INTERVENTIONS:
Device: Selective Retina Therapy (SRT) — SRT (pulsed double-Q-switched Nd-YLF laser, wavelength 527 nm, t=1.7 µs, energy 100-370 μJ).
  Other Names: SRT-Laser system (Medical Laser Center Lübeck, Germany)
  Arms: Selective Retinatherapy (SRT); crossover

SUMMARY:
The purpose of this study is to evaluate the efficacy of Selective Retina Therapy (SRT) for treating acute idiopathic central serous chorioretinopathy (ICSC). Patients with acute symptomatic ICSC of at least 3 months duration were recruited. The patients were randomized by equal terms to SRT- (Treatment) and control group. After 3 months follow up patients of control group with persistence of disease activity were allocated to crossover group and received either SRT. Crossover group was followed up for further 3 months.

The primary outcome measure of the study are the serial changes in Early Treatment of Diabetic Retinopathy Study (ETDRS) letterscore and edema in optical coherence tomography (OCT) at 3 months. Secondary outcome measures included the proportion of eyes with complete absorption of subretinal fluid, leakage in fluorescein angiography and the systemic and ocular complications during the study at 3 months.

DETAILED DESCRIPTION:
Idiopathic central serous chorioretinopathy (ICSC) is characterized by a serous detachment of the neurosensory retina in the macular region secondary to a focal or retinal pigment epithelial defect. Patients with ICSC, oftentimes young male adults, experience visual disturbances including micropsia, metamorphopsia, central scotoma, reduced visual acuity and loss of contrast sensitivity. Most cases of ICSC are presumed to be self-limiting and usually resolve spontaneously within 3 to 4 months.Nevertheless the duration of the disease is strongly related to the vision prognosis and reattachment within 4 months of onset is considered as a relevant therapeutic target because prolonged detachment is associated with photoreceptor atrophy.

The therapeutic effect of focal cw laser photocoagulation has not been fully established. One obvious theory postulates that the beneficial effect of photocoagulation is associated with the establishment of a new barrier of RPE cells which subsequently reintegrate the RPE pump function and the integrity of the RPE as a barrier. Based on this theory, the destruction of tissues surrounding the RPE, in particular Bruch's membrane, the choroid and the photoreceptors, would be an unwanted side effect. On the basis of this consideration Selective Retina Therapy (SRT), which is a innovative laser technology that selectively damages the RPE and spares the neurosensory retina, suggests itself as an ideal treatment for ICSC with focal leakage, especially if the RPE leak is located close to the fovea.

It has been proved as safe, and microperimetry has shown that SRT does not cause microscotoma. SRT has already been adopted in the treatment of diverse macular diseases inter alia in patients with ICSC with promising performance.

ELIGIBILITY:
Inclusion Criteria:

* Anamnestic reduction of visual acuity
* Atients with best-corrected visual acuity (BCVA) of 20/200 or better
* Presence of subretinal fluid (SRF) on optical coherence tomography (OCT)
* Presence of active angiographic (multi)focal leakage in fluorescein angiography (FA) caused by ICSC but not choroidal neovascularisation (CNV) or other diseases
* Absence of other retinal or ocular diseases (e. g. glaucoma, vessel diseases, vein occlusion or proliferative retinopathy)
* Absence of cataract or media opacities of a degree which precludes taking retinal photographs and FA's
* Absence of angle closure glaucoma which precludes pharmacological dilatation of the pupil.

Exclusion Criteria:

* Patients who received any previous treatment, including PDT or focal cw laser photocoagulation for ICSC, or who had evidence of CNV, PCV, or other maculopathy on clinical examination or FA were excluded.
* Patients receiving exogenous corticosteroid treatment, with systemic diseases such as Cushing's disease or renal diseases, and pregnant patients also were excluded.
* Informed consent was obtained from all subjects, and the study protocol was approved by the ethics committee of the University of Kiel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Serial changes in ETDRS letterscore | 3 months

SECONDARY OUTCOMES:
The maximum distance between the RPE and the outer neurosensory retina in the area of Subretinal fluid accumulation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Johann J Roider, Professor, Study Director — Department of Ophthalmology University of Kiel
Locations (1):
- Department of Ophthalmology, Kiel, Schleswig-Holstein, Germany

REFERENCES:
- [Result] Elsner H, Porksen E, Klatt C, Bunse A, Theisen-Kunde D, Brinkmann R, Birngruber R, Laqua H, Roider J. Selective retina therapy in patients with central serous chorioretinopathy. Graefes Arch Clin Exp Ophthalmol. 2006 Dec;244(12):1638-45. doi: 10.1007/s00417-006-0368-5. PMID 16758179
- [Result] Klatt C, Elsner H, Porksen E, Brinkmann R, Bunse A, Birngruber R, Roider J. [Selective retina therapy in central serous chorioretinopathy with detachment of the pigmentary epithelium]. Ophthalmologe. 2006 Oct;103(10):850-5. doi: 10.1007/s00347-006-1415-7. German. PMID 16937094
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203
- [Derived] Klatt C, Saeger M, Oppermann T, Porksen E, Treumer F, Hillenkamp J, Fritzer E, Brinkmann R, Birngruber R, Roider J. Selective retina therapy for acute central serous chorioretinopathy. Br J Ophthalmol. 2011 Jan;95(1):83-8. doi: 10.1136/bjo.2009.178327. Epub 2010 Jun 15. PMID 20554506
- See also: homepage of the Medical Laser Center Lübeck, Lübeck, Germany. — http://www.mll-luebeck.de/admin/srt.htm